CLINICAL TRIAL: NCT06115070
Title: Intravenous Thrombolytic Therapy for Acute Ischemic Stroke Patients with Low NIHSS and Non-disabling Deficits
Acronym: ALLOW
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ALLOW
Record Dates: First submitted 2023-10-19; First posted 2023-11-02 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-02

CONDITIONS: Thrombosis; Acute Ischemic Stroke (AIS)
MeSH Terms: conditions — Thrombosis; Ischemic Stroke | interventions — Tissue Plasminogen Activator

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intravenous thrombolysis (alteplase and other guideline-recommended thrombolytic agents) (Experimental): Patients will receive standard dose intravenous alteplase (0.9 mg/kg, the first 10% administered as an initial bolus and the remainder over a 1-hour period, with a maximum dose of 90 mg)，intravenous Tenecteplase(0.25mg/kg，administered as a single intravenous bolus injection over 5 - 10 seconds，with a maximum dose of 25 mg), intravenous reteplase (a bolus of 18 mg followed by a second bolus of 18 mg after 30 minutes) and intravenous prourokinase (rhPro-UK) (15 mg bolus followed by a 20 mg infusion over 30 minutes).
  Interventions: Drug: Intravenous thrombolysis (alteplase and other guideline-recommended thrombolytic agents)
- Standard therapy (No Intervention): Standard therapy

INTERVENTIONS:
Drug: Intravenous thrombolysis (alteplase and other guideline-recommended thrombolytic agents) — Patients will receive standard dose intravenous alteplase (0.9 mg/kg, the first 10% administered as an initial bolus and the remainder over a 1-hour period, with a maximum dose of 90 mg)，intravenous Tenecteplase(0.25mg/kg，administered as a single intravenous bolus injection over 5 - 10 seconds，with a maximum dose of 25 mg), intravenous reteplase (a bolus of 18 mg followed by a second bolus of 18 mg after 30 minutes) and intravenous prourokinase (rhPro-UK) (15 mg bolus followed by a 20 mg infusion over 30 minutes).
  Arms: Intravenous thrombolysis (alteplase and other guideline-recommended thrombolytic agents)

SUMMARY:
Minor stroke is considered an acute ischemic stroke (AIS) that has a National Institute of Health Stroke Scale (NIHSS) score ≤ 5 points. About 1/3 patients with mild stroke have poor prognosis, whether patients with this type undergo thrombolysis has been a controversial issue. A pooled analysis published in the Lancet in 2014 included 9 high-quality RCT studies of intravenous thrombolysis such as NINDS and IST3, and a total of 666 (10%) patients with mild stroke were included in the analysis. For mild stroke, the proportion of good prognosis in the control group and the alteplase group was 58.9% and 68.7% (OR 1.48, 95%Cl 1.07-2.06), respectively. Therefore, guidelines recommended alteplase thrombolytic therapy for patients with mild stroke. However, PRISMS, a randomized controlled trial of intravenous thrombolytic therapy for mild stroke published in 2018, found that alteplase intravenous thrombolytic therapy did not improve clinical outcomes compared with aspirin in patients with mild non-disabled stroke (90-day mRS 0-1 ratio 78.2% vs 81.5%), and the incidence of symptomatic intracranial hemorrhage was higher. However, a major limitation of the PRISMS study was that more than 85% of patients had numbness and dysarticulation, so this conclusion cannot be extrapolated to patients with other mild stroke symptoms. Moreover, due to the early termination of the sponsorship of this trial, the number of enrolled cases did not reach the pre-designed number, resulting in a serious decline in the authenticity of the study results. Symptoms and outcomes of minor stroke are important criteria for assessment. However, there is currently no uniform standard for the assessment of disability.

Both international and domestic guidelines recommend IVT with alteplase for minor disabling stroke within 4.5h, but not routinely recommend intravenous thrombolysis for minor nondisabling stroke within 4.5h. It is important to underline that strokes with low NIHSS scores are not necessarily nondisabling. Despite, patients with mild stroke symptoms are often excluded from IVT due to safety concerns potentially outweighing the putative benefits of recanalization therapy.

Therefore, the investigators developed a new definition to refine the disability assessment of stroke symptoms. The purpose of this study was to investigate whether AIS patients with NIHSS ≤ 5, a limb-related NIHSS item score of 0, and with any of the following NIHSS item ≥2: Best Gaze, Visual, Facial palsy, Limb ataxia, Sensory, Best language, Dysarthria, Extinction and Inattention, could benefit from intravenous thrombolysis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with clinical signs of acute ischemic stroke within 4.5 hours of onset or awakening with stroke (if within 4.5 hours from the midpoint of sleep).
2. Patinet's age is >18 years
3. Patients with NIHSS ≤ 5, a limb-related NIHSS item score of 0, and with any of the following NIHSS item ≥2: Best Gaze, Visual, Facial palsy, Limb ataxia, Sensory, Best language, Dysarthria, Extinction and Inattention.

Exclusion Criteria:

(1) Plan to receive endovascular treatment; (2) Pre-stroke mRS score > 2 (3) Contraindications for IVT：

1. Intracranial hemorrhage (including parenchymal hemorrhage, intraventricular hemorrhage, subarachnoid hemorrhage, epidural hematoma, etc.)
2. Previous history of intracranial hemorrhage
3. Severe head trauma or stroke history within the last 3 months
4. Intracranial tumors, giant intracranial aneurysms
5. Intracranial or spinal surgery within the recent 3 months
6. Major surgical procedures within the last 2 weeks
7. Gastrointestinal or urinary tract bleeding within the last 3 weeks
8. Active visceral bleeding
9. Aortic arch dissection
10. Arterial puncture in a site within the last 1 week that is not easy to compress and stop bleeding
11. Elevated blood pressure: Systolic blood pressure ≥ 180 mmHg or diastolic blood pressure ≥ 100 mmHg
12. Acute bleeding tendency, including platelet count < 100 × 10⁹/L or other conditions
13. Received low-molecular-weight heparin treatment within 24 hours
14. Oral anticoagulants (warfarin) with INR > 1.7 or PT > 15 s; Receiving heparin treatment with aPTT above the upper limit of the normal range within the last 24 hours of onset, Receiving thrombin inhibitors and factor Xa inhibitors within the last 48 hours of onset.
15. Blood sugar < 2.8 or > 22.22 mmol/L
16. Head CT or MRI indicates large-area infarction (infarction area ≥ 1/3 of the middle cerebral artery supply area) (4) The judgment is left to the discretion of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 390 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Excellent recovery assessed by the ratio of modified Rankin Scale (mRS) score of 0-1 (%) at 90 ± 7 days | 90 ± 7 days
  mRS: minimum value = 0, maximum value = 6, and lower scores mean a better outcome

SECONDARY OUTCOMES:
Independent recovery assessed by ratio of modefied Rankin Scale (mRS) score of 0-2 (%) at 90 ± 7 days | 90 ± 7 days
  mRS: minimum value = 0, maximum value = 6, and lower scores mean a better outcome
recovery assessed by modefied Rankin Scale (mRS) score | 90 ± 7 days
  mRS: minimum value = 0, maximum value = 6, and lower scores mean a better outcome
3-month mortality | 90 ± 7 days
  Hospitalization records or follow-up results
the change on the NIHSS score from baseline to 24 hours | 24 hours
  NIHSS: minimum value = 0, maximum value = 42, and higher scores mean severer symptoms
Presence of hemorrhagic transformation evaluated by CT or MRI | at day 1
  Presence of hemorrhagic transformation is defined according the standard from ECASS-2 study
Presence of parenchymal hemorrhage (PH) evaluated by CT or MRI | at day 1
  the presence of PH is defined according the standard from ECASS-2 study
Presence of symptomatic intracerebral hemorrhage (sICH) evaluated by CT or MRI | at day 1
  the presence of sICH is defined according the standard from ECASS-2 study

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affiliated Hospital of Zhejiang University, School of Medicine, Hangzhou, China

IPD SHARING:
Plan to Share IPD: No